CLINICAL TRIAL: NCT01799382
Title: Mutational Analysis of Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA) Specimens in Patients With Advanced Non-small Cell Lung Cancer: a Randomized Trial of Rapid On-site Evaluation
Brief Title: Role of Rapid On-site Evaluation for Mutational Analysis of EBUS-TBNA Specimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Rocco Trisolini, M.D., Maggiore Bellaria Hospital, Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13001-Trisolini
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Rapid On-site Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA + Rapid on-site evaluation (Experimental): Patients in this arm will undergo rapid-on site evaluation of samples obtained with EBUS-TBNA
  Interventions: Other: Rapid on-site evaluation; Device: EBUS-TBNA
- EBUS-TBNA (Active Comparator): Patients in this arm will undergo EBUS-TBNA without rapid on-site evaluation
  Interventions: Device: EBUS-TBNA

INTERVENTIONS:
Other: Rapid on-site evaluation — Rapid on-site evaluation consists on the cytological evaluation of samples obtained during a diagnostic procedure by a pathologist present in the diagnostic suite. In the present study, cytological samples obtained with EBUS-TBNA during bronchoscopy will be evaluated.
  Arms: EBUS-TBNA + Rapid on-site evaluation
Device: EBUS-TBNA — EBUS-TBNA is a needle aspiration procedure guided by endobronchial ultrasounds performed during bronchoscopy

SUMMARY:
The purpose of the study is to determine if rapid on-site evaluation of EBUS-TBNA samples can increase the percentage of patients with advanced non-squamous non-small cell lung cancer in whom both pathologic subtyping and mutational analysis are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Suspected hilar or mediastinal lymph node metastasis from lung cancer

Exclusion Criteria:

* Pregnancy
* Uncontrolled coagulopathy
* Refusal to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mutational analysis of epidermal growth factor receptor (EGFR), K-ras, and ALK (anaplastic lymphoma kinase) genes | 18 months
  Percentage of patients for whom the mutational analysis of epidermal growth factor receptor (EGFR), K-ras, and ALK (anaplastic lymphoma kinase) genes on EBUS-TBNA samples is obtained

SECONDARY OUTCOMES:
Diagnostic yield of EBUS-TBNA | 18 months
Adequacy of EBUS-TBNA samples | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Maggiore Hospital, Bologna, Italy
Locations (1):
- Maggiore Hospital, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Derived] Trisolini R, Cancellieri A, Tinelli C, de Biase D, Valentini I, Casadei G, Paioli D, Ferrari F, Gordini G, Patelli M, Tallini G. Randomized Trial of Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration With and Without Rapid On-site Evaluation for Lung Cancer Genotyping. Chest. 2015 Dec;148(6):1430-1437. doi: 10.1378/chest.15-0583. PMID 26158441